CLINICAL TRIAL: NCT07094048
Title: Immunoglobulins in Multiple Myeloma Patients Receiving a BCMA-Directed T Cell Engager
Acronym: CHUQUL_HO001
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MP-20-2025-7948
Record Dates: First submitted 2025-07-11; First posted 2025-07-30 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma Refractory; Relapsed Multiple Myeloma
Keywords: Immunoglobulins; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Standard of Care; Crossing Over, Genetic

STUDY DESIGN:
Intervention Model Description: Of note, patients in Group C will crossover to Group A or B once meeting the pre specified conditions.
  Stratified randomization with block design by site.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A IgG level 8-10 g/L (Active Comparator): Immunoglobulin support (subcutaneous or intravenous)
  Interventions: Drug: Target trough IgG level of 8-10 g/L
- Group B IgG level 4-6 g/L (Experimental): Immunglobulin support (subcutaneous or intravenous)
  Interventions: Drug: Target trough IgG level 4-6 g/L
- Group C (Other): No immunoglobulin support. If pre specified conditions are met, crossover to Group A or B.
  Interventions: Drug: No history of recurrent or severe infections and total IgG level higher or equal at 4 g/L

INTERVENTIONS:
Drug: Target trough IgG level of 8-10 g/L — Target trough IgG level of 8-10 g/L
  Other Names: Standard of care
  Arms: Group A IgG level 8-10 g/L
Drug: Target trough IgG level 4-6 g/L — Target trough IgG level of 4-6 g/L
  Other Names: Experimental
  Arms: Group B IgG level 4-6 g/L
Drug: No history of recurrent or severe infections and total IgG level higher or equal at 4 g/L — If, during follow-up, the patient presents recurrent or severe infections and/or total IgG level less 4 g/L, crossover to group A or B
  Other Names: Crossover
  Arms: Group C

SUMMARY:
Bispecific antibody therapies targeting BCMA (B-cell maturation antigen) represent a novel therapeutic approach for patients with multiple myeloma. They are currently used in cases of refractory multiple myeloma but are also being investigated in earlier lines of treatment. However, these new therapies can lead to deeper immunosuppression and exacerbate an underlying immunosuppressive state in patients with multiple myeloma. As a result, infectious complications are common with these therapies and are a significant concern. Therefore, preventing infections in this population is crucial. However, data on the best strategies for prevention are currently lacking.

DETAILED DESCRIPTION:
Although the effectiveness of immunoglobulins (Ig) has been demonstrated, it remains to be determined whether immunoglobulin administration is necessary for all patients receiving these therapies or only for those with low serum immunoglobulin G (IgG) levels. Furthermore, the optimal target IgG level to achieve in order to reduce the risk of infections is also unknown in this specific population of multiple myeloma patients. Guidance needs to be provided to the clinicians to better support MM patients undergoing this novel therapy by addressing the hypogammaglobulinemia and therefore limiting and ideally avoiding the high risk of infections.

In this prospective, randomized, unblinded, multicenter study, as per the standard of care approach, every patient with relapsed refractory MM receiving a BCMA-directed TCE with history of recurrent or severe infections and/or total IgG level less than 4 g/L will receive Ig support (intravenous ou subcutaneous). Once on Ig supplementation, the optimal target trough IgG level to achieve is not well established. The goal of this study is therefore to better define, in this patient population , the target trough IgG level to achieve a reduction in the incidence of severe infections.

The primary objective is to demonstrate the non-inferiority in the cumulative incidence of severe infections at 3 months between patients on Ig support with a target trough IgG level of 4-6 g/L (experimental group) versus a target trough IgG level of 8-10 g/L (standard of care (SOC) group).

ELIGIBILITY:
Inclusion Criteria:

* Multiple myeloma patient:
* ≥ 18 years old
* ≥ 1 prior lines of therapy
* Receiving a BCMA-directed T-cell Engager therapy (starting on treatment)
* On previous Ig support or not

Exclusion Criteria:

* Less than 18 years old
* Pregancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Severe infections | From enrollment to 3 months after time of randomization
  Non-inferiority in the cumulative incidence of severe infections at 3 months between patients on Ig support with a target trough IgG level of 4-6 g/L (experimental group) versus a target trough IgG level of 8-10 g/L (standard of care group)

SECONDARY OUTCOMES:
Minor/Moderate infections rate | From enrollment to 12 monts after randomization
  Rates of minor/moderate infection rates
All infection rate | From enrollment to 12 months after randomization
  All infections rate

OTHER OUTCOMES:
Vaccinal response (optional) | From vaccination (at enrollment) to 1 month after vaccination.
  For patients with no previous Ig support, we will examine the vaccinal response with specific antibody titers to tetanus.
CM reactivation and infection rate | From enrollment to 12 months after randomization
  CMV reactivation and infection
Adverse events related to the administration of the Ig product | From enrollment to 12 months after randomization
  Adverse events related to the administration of the Ig product
Quality of life assessment, according to the EORTC-QLQ-C30 | From enrollment to 12 months after randomization
  Quality of life assessment (SC and IV)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Julie Côté, MD,FRCPC, Study Chair — CHU de Québec-Université Laval; Dr Julie Côté, MD,FRCPC, Principal Investigator — CHU de Québec-Université Laval; Dr Vincent Laroche, MD,FRCPC, Principal Investigator — CHU de Québec-Université Laval
Locations (1):
- Centre Intégré de Cancérologie, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mohan M, Monge J, Shah N, Luan D, Forsberg M, Bhatlapenumarthi V, Balev M, Patwari A, Cheruvalath H, Bhutani D, Thanendrarajan S, Dhakal B, Zangari M, Al-Hadidi S, Cooper D, Lentzsch S, van Rhee F, D'Souza A, Szabo A, Schinke C, Chakraborty R. Teclistamab in relapsed refractory multiple myeloma: multi-institutional real-world study. Blood Cancer J. 2024 Mar 5;14(1):35. doi: 10.1038/s41408-024-01003-z. PMID 38443345
- [Background] Compagno N, Cinetto F, Semenzato G, Agostini C. Subcutaneous immunoglobulin in lymphoproliferative disorders and rituximab-related secondary hypogammaglobulinemia: a single-center experience in 61 patients. Haematologica. 2014 Jun;99(6):1101-6. doi: 10.3324/haematol.2013.101261. Epub 2014 Mar 28. PMID 24682509
- [Background] Gardulf A, Nicolay U, Math D, Asensio O, Bernatowska E, Bock A, Costa-Carvalho BT, Granert C, Haag S, Hernandez D, Kiessling P, Kus J, Matamoros N, Niehues T, Schmidt S, Schulze I, Borte M. Children and adults with primary antibody deficiencies gain quality of life by subcutaneous IgG self-infusions at home. J Allergy Clin Immunol. 2004 Oct;114(4):936-42. doi: 10.1016/j.jaci.2004.06.053. PMID 15480339
- [Background] Ducruet T, Levasseur MC, Des Roches A, Kafal A, Dicaire R, Haddad E. Pharmacoeconomic advantages of subcutaneous versus intravenous immunoglobulin treatment in a Canadian pediatric center. J Allergy Clin Immunol. 2013 Feb;131(2):585-7.e1-3. doi: 10.1016/j.jaci.2012.08.022. Epub 2012 Oct 2. No abstract available. PMID 23040368
- [Background] Martin A, Lavoie L, Goetghebeur M, Schellenberg R. Economic benefits of subcutaneous rapid push versus intravenous immunoglobulin infusion therapy in adult patients with primary immune deficiency. Transfus Med. 2013 Feb;23(1):55-60. doi: 10.1111/j.1365-3148.2012.01201.x. Epub 2012 Nov 20. PMID 23167310
- [Background] Perez EE, Orange JS, Bonilla F, Chinen J, Chinn IK, Dorsey M, El-Gamal Y, Harville TO, Hossny E, Mazer B, Nelson R, Secord E, Jordan SC, Stiehm ER, Vo AA, Ballow M. Update on the use of immunoglobulin in human disease: A review of evidence. J Allergy Clin Immunol. 2017 Mar;139(3S):S1-S46. doi: 10.1016/j.jaci.2016.09.023. Epub 2016 Dec 29. PMID 28041678
- [Background] Gardulf A. Immunoglobulin treatment for primary antibody deficiencies: advantages of the subcutaneous route. BioDrugs. 2007;21(2):105-16. doi: 10.2165/00063030-200721020-00005. PMID 17402794
- [Background] Stiehm ER. Adverse effects of human immunoglobulin therapy. Transfus Med Rev. 2013 Jul;27(3):171-8. doi: 10.1016/j.tmrv.2013.05.004. Epub 2013 Jul 6. PMID 23835249
- [Background] Jolles S, Michallet M, Agostini C, Albert MH, Edgar D, Ria R, Trentin L, Levy V. Treating secondary antibody deficiency in patients with haematological malignancy: European expert consensus. Eur J Haematol. 2021 Apr;106(4):439-449. doi: 10.1111/ejh.13580. Epub 2021 Feb 2. PMID 33453130
- [Background] Otani IM, Lehman HK, Jongco AM, Tsao LR, Azar AE, Tarrant TK, Engel E, Walter JE, Truong TQ, Khan DA, Ballow M, Cunningham-Rundles C, Lu H, Kwan M, Barmettler S. Practical guidance for the diagnosis and management of secondary hypogammaglobulinemia: A Work Group Report of the AAAAI Primary Immunodeficiency and Altered Immune Response Committees. J Allergy Clin Immunol. 2022 May;149(5):1525-1560. doi: 10.1016/j.jaci.2022.01.025. Epub 2022 Feb 14. PMID 35176351
- [Background] Guo Y, Tian X, Wang X, Xiao Z. Adverse Effects of Immunoglobulin Therapy. Front Immunol. 2018 Jun 8;9:1299. doi: 10.3389/fimmu.2018.01299. eCollection 2018. PMID 29951056
- [Background] Orange JS, Grossman WJ, Navickis RJ, Wilkes MM. Impact of trough IgG on pneumonia incidence in primary immunodeficiency: A meta-analysis of clinical studies. Clin Immunol. 2010 Oct;137(1):21-30. doi: 10.1016/j.clim.2010.06.012. Epub 2010 Aug 1. PMID 20675197
- [Background] Lee JL, Mohamed Shah N, Makmor-Bakry M, Islahudin FH, Alias H, Noh LM, Mohd Saffian S. A Systematic Review and Meta-regression Analysis on the Impact of Increasing IgG Trough Level on Infection Rates in Primary Immunodeficiency Patients on Intravenous IgG Therapy. J Clin Immunol. 2020 Jul;40(5):682-698. doi: 10.1007/s10875-020-00788-5. Epub 2020 May 16. PMID 32417999
- [Background] Raje N, Anderson K, Einsele H, Efebera Y, Gay F, Hammond SP, Lesokhin AM, Lonial S, Ludwig H, Moreau P, Patel K, Ramasamy K, Mateos MV. Monitoring, prophylaxis, and treatment of infections in patients with MM receiving bispecific antibody therapy: consensus recommendations from an expert panel. Blood Cancer J. 2023 Aug 1;13(1):116. doi: 10.1038/s41408-023-00879-7. PMID 37528088
- [Background] Frerichs KA, Verkleij CPM, Mateos MV, Martin TG, Rodriguez C, Nooka A, Banerjee A, Chastain K, Perales-Puchalt A, Stephenson T, Uhlar C, Kobos R, van der Holt B, Kruyswijk S, Kuipers MT, Groen K, Vishwamitra D, Skerget S, Cortes-Selva D, Doyle M, Zaaijer HL, Zweegman S, Verona RI, van de Donk NWCJ. Teclistamab impairs humoral immunity in patients with heavily pretreated myeloma: importance of immunoglobulin supplementation. Blood Adv. 2024 Jan 9;8(1):194-206. doi: 10.1182/bloodadvances.2023011658. PMID 38052042
- [Background] Lancman G, Parsa K, Kotlarz K, Avery L, Lurie A, Lieberman-Cribbin A, Cho HJ, Parekh SS, Richard S, Richter J, Rodriguez C, Rossi A, Sanchez LJ, Thibaud S, Jagannath S, Chari A. IVIg Use Associated with Ten-Fold Reduction of Serious Infections in Multiple Myeloma Patients Treated with Anti-BCMA Bispecific Antibodies. Blood Cancer Discov. 2023 Nov 1;4(6):440-451. doi: 10.1158/2643-3230.BCD-23-0049. PMID 37769148
- [Background] Lesokhin AM, Tomasson MH, Arnulf B, Bahlis NJ, Miles Prince H, Niesvizky R, Rodriotaguez-Otero P, Martinez-Lopez J, Koehne G, Touzeau C, Jethava Y, Quach H, Depaus J, Yokoyama H, Gabayan AE, Stevens DA, Nooka AK, Manier S, Raje N, Iida S, Raab MS, Searle E, Leip E, Sullivan ST, Conte U, Elmeliegy M, Czibere A, Viqueira A, Mohty M. Elranatamab in relapsed or refractory multiple myeloma: phase 2 MagnetisMM-3 trial results. Nat Med. 2023 Sep;29(9):2259-2267. doi: 10.1038/s41591-023-02528-9. Epub 2023 Aug 15. PMID 37582952
- [Background] Moreau P, Garfall AL, van de Donk NWCJ, Nahi H, San-Miguel JF, Oriol A, Nooka AK, Martin T, Rosinol L, Chari A, Karlin L, Benboubker L, Mateos MV, Bahlis N, Popat R, Besemer B, Martinez-Lopez J, Sidana S, Delforge M, Pei L, Trancucci D, Verona R, Girgis S, Lin SXW, Olyslager Y, Jaffe M, Uhlar C, Stephenson T, Van Rampelbergh R, Banerjee A, Goldberg JD, Kobos R, Krishnan A, Usmani SZ. Teclistamab in Relapsed or Refractory Multiple Myeloma. N Engl J Med. 2022 Aug 11;387(6):495-505. doi: 10.1056/NEJMoa2203478. Epub 2022 Jun 5. PMID 35661166